CLINICAL TRIAL: NCT04744038
Title: Evaluating the Efficacy of Positive Airway Pressure Therapy for Treating Obstructive Sleep Apnea in the Home Environment
Brief Title: Evaluating the Efficacy of PAP Therapy for Treating OSA in the Home Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLP-20-01-01
Record Dates: First submitted 2021-01-04; First posted 2021-02-08 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Investigational Device (Experimental): Participants will then be asked to take home the investigational device to use at night while they sleep in place of their own device. The participant's therapy and comfort settings will be copied from their own device to the investigational device. Participants will use their own mask with the investigational device for the duration of this study.
  Interventions: Device: Positive Airway Pressure (PAP) Therapy

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) Therapy — PAP therapy supplies pressurized air from the flow generator to the upper airway via air tubing and a mask to prevent the repetitive collapse of the upper airway during sleep.

SUMMARY:
This study will take between 4-6 months (with first patient first visit to last patient last visit expected to span 3-4 months across all study sites). Each participant will use the investigational PAP device with their own mask for a period of up to 7 nights and will complete a series of questionnaires upon completion. The study will evaluate the usability and efficacy of the investigational device in the intended use environment by the intended use population.

DETAILED DESCRIPTION:
A new PAP device has been developed by ResMed which includes an improved humidification system, a new user interface and optimized workflows. This study will assess the efficacy and usability of the new PAP device in an OSA population.

This is a prospective, open-label, single arm study, multi-site study to assess the usability and efficacy of investigational device in the home environment.

Recruitment Recruitment will be done via phone calls/ SMS messages/ emails. Participants will be explained the details of the study and those who wish to take part will be invited to a ResMed clinic or selected site for the first study visit (As detailed in section 7).

Visit 1 Participants will provide written informed consent (as per section 6.1). If eligible, baseline participant demographics will be collected. Participants will be shown the investigation device. If the participant is happy to proceed the investigational device will be set-up to be exactly the same as their current CPAP device, and the participant will take it home to use in place of their own device.

Visit 2 At the conclusion of the 7 nights of use, the participant will be asked to fill in a questionnaire documenting their experience with the investigational device. The participant will return all study equipment to the researcher. The questionnaires will be reviewed. This concludes the participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients who ≥ 18 years of age
* Patients being established on PAP therapy for the treatment of OSA for ≥ 6 months
* Patients currently using AirSense10 (as their primary device)
* Patients currently using an appropriate mask system (AirFit F20, AirFit P10, AirFit N20, AirFit N30i, AirFit F30i or AirFit P30i)
* Patients who can trial the investigational device for up to 7 nights
* Patients who have been compliant to therapy (average of ≥4 hours of usage) for the previous 7 nights of use* *the most recent consecutive 7 nights within the last 30 days

Exclusion Criteria:

* Patients using Bilevel flow generators
* Patients who are or may be pregnant
* Patients with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Patients believed to be unsuitable for inclusion by the researcher
* Patients who or whose bed partner has implantable metallic implants in the head, neck and chest region affected by magnetic fields (Non-ferrous implants may be acceptable)
* Patients using supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Usability | 1 week
  Subjective ratings of the Usability of the Pacific device after using it in the home environment for up to 7 nights. Ratings will be collected using an 11 point Likert Scale where a score of 10 is considered very favorable, and a score of 0 is very unfavorable.

SECONDARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 1 week
  Number of residual Apnea Hypopnea events within a clinically acceptable range when using the Pacific device in the home environment for a up to 7 nights.
Usage-Positive Airway Pressure (PAP) Device parameters | 1 week
  Average number of hours per night of use of the Pacific Device during sleep sessions from up to 7 nights
Leak-Positive Airway Pressure (PAP) Device parameters | 1 week
  Average median, 95 percentile and maximum leak(L/min) while using the Pacific device from up to 7 nights
Pressure-Positive Airway Pressure (PAP) Device parameters | 1 week
  Average pressure delivered by the Pacific device between 4cmH2O-20cmH2O from use up to 7 nights
Acoustic Signals | 1 week
  Cross-correlation of the acoustic signals recorded from the patient environment and the external recording in the controlled laboratory environment identification algorithm.

CONTACTS AND LOCATIONS:
Locations (2):
- Sleep Data, San Diego, California, United States
- ResMed BELLA VISTA, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No